CLINICAL TRIAL: NCT01885442
Title: TryCYCLE (Critical Care Cycling to Improve Lower Extremity Strength): A Prospective Pilot Study of the Safety and Feasibility of Early In-bed Leg Cycle Ergometry in Mechanically Ventilated Patients
Brief Title: TryCYCLE: A Pilot Study of Early In-bed Leg Cycle Ergometry in Mechanically Ventilated Patients
Acronym: TryCYCLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TryCYCLE
Record Dates: First submitted 2013-03-21; First posted 2013-06-25 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Intensive Care Unit Acquired Weakness; Critical Care; Mechanical Ventilation; Respiratory Failure
Keywords: mechanical ventilation; cycle ergometry; intensive care unit; rehabilitation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- In-bed leg cycle ergometry (Experimental)
  Interventions: Device: In-bed leg cycle ergometry

INTERVENTIONS:
Device: In-bed leg cycle ergometry — Patients will receive 30 minutes of in-bed leg cycling in addition to routine physiotherapy, 6 days per week, for the duration of their ICU stay (to a maximum of 28 days).
  Other Names: RT300 Supine Cycle Ergometer (Restorative Therapies, Baltimore, MD)

SUMMARY:
Background: Patients in the intensive care unit (ICU) are the sickest in hospital, and need advanced life-support. Survivors of critical illness are very vulnerable to weakness and disability. Up to 1 in 4 have severe leg weakness impairing their quality of life for as long as 5 years after ICU discharge. In-bed cycling employs special equipment that attaches to a patient's hospital bed, allowing them gentle leg exercise while in the ICU. The investigators will offer patients in-bed cycling while they are needing a breathing machine, to help them recover from weakness as fast as possible. Before doing a larger trial testing if in-bed cycling reduces disability, data on safety (Is it safe?) and feasibility (Can the investigators do it?) are needed.

Objectives: To study the safety and feasibility of in-bed leg cycling in critically ill patients who need breathing machines.

Methods: Adult patients admitted to the ICU who need a breathing machine and are expected to survive their ICU stay are eligible. Specially trained physiotherapists will provide patients with 30 minutes of in-bed cycling each day while they are in the ICU.

Outcomes: The investigators will study (1) Safety: the heart rate and breathing patterns of patients doing in-bed cycling, while carefully monitoring for safety. (2) Feasibility: whether patients can cycle on most days of their ICU stay, whether patients and their families agree to be a part of the study, and whether the investigators can assess patients' strength in the ICU and at hospital discharge.

Relevance: As the Canadian population ages, the demand for breathing machines during acute illness will increase dramatically. Effective methods of physiotherapy are needed for critically ill patients to minimize muscle weakness, speed recovery, and improve quality of life. This pilot study is the first of several future larger studies about in-bed cycling in the ICU. This program of research will help patients needing life support to regain their strength and recover as fast as possible from critical illness.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years old
* Invasively mechanically ventilated ≤4 days
* Expected additional 2 day ICU stay
* Ability to ambulate independently pre-hospital (with or without a gait aid)

Exclusion Criteria:

* Unable to follow simple commands at baseline
* Pregnancy
* Acute conditions impairing ability to walk or cycle (e.g., leg or foot fracture)
* Acute central condition or peripheral injury resulting in neuromuscular weakness (e.g., stroke, Guillain Barré syndrome)
* Primary generalized weakness of the central or peripheral nervous system (e.g., multiple sclerosis, myasthenia gravis, Parkinson's disease, amyotrophic lateral sclerosis)
* Temporary pacemaker wires
* Expected hospital mortality> 90%
* Cycling equipment unable to fit patient's body dimensions (e.g., leg amputation or obesity)
* Specific surgical exclusion as stipulated by attending

  ->7 day ICU stay
* Physician declines
* Patient did not meet daily screening criteria to provide in-bed leg cycling during the first 4 days of mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of in-bed leg cycling research sessions terminated (composite outcome) | From date of enrollment until date of ICU discharge, approximately 10 days on average
  Research sessions will stop if the patient meets any of the following criteria:
  * Sustained oxygen desaturation <88%, despite adjustments to FiO2
  * Heart rate
    * Low: 20 bpm less than lowest baseline value or 40 bpm (whichever is highest)
    * High: 20 bpm more than highest baseline value or 140 bpm (whichever is lowest)
  * Mean Arterial Pressure <55 or >110 mmHg
  * Marked ventilator dyssynchrony not corrected by adjusting cycle off criteria
  Safety events:
  * Suspected new unstable / uncontrolled arrhythmia
  * Concern for myocardial ischaemia
  * Respiratory distress leading to symptoms of intolerable dyspnea
  * Unplanned extubation Any of the following catheter or tube dislodgements
  * Catheters: Central venous, arterial, dialysis, or pulmonary artery catheter
  * Tubes: Orogastric, nasogastric, or percutaneous endoscopic gastrostomy
  ICU physician, patient or proxy requests termination of session

SECONDARY OUTCOMES:
Number of adverse events: Intravascular catheter or tube dislodgement rate during in-bed cycling | From date of enrollment until date of ICU discharge, approximately 10 days on average
  Any of the following catheter or tube dislodgements:
  * Catheters: Central venous, arterial, dialysis, or pulmonary artery catheter
  * Tubes: Orogastric, nasogastric, or percutaneous endoscopic gastrostomy
Daily research session delivery rate | From date of enrollment until date of ICU discharge, approximately 10 days on average
  We will assess our ability to deliver cycling during the ICU stay by comparing our daily delivery rate with that achieved in ICU rehabilitation randomized clinical trials (80%).
Rate of outcome measure ascertainment in assessable patients at ICU awakening | 5 days after study admission, on average
  We will calculate the binary proportion and 95% confidence interval for outcome measure ascertainment event rates.
Rate of outcome measure ascertainment in assessable patients at ICU discharge | 10 days after study admission, on average
  We will calculate the binary proportion and 95% confidence interval for outcome measure ascertainment event rates.
Rate of outcome measure ascertainment in assessable patients at hospital discharge | 15 days after study admission, on average
  We will calculate the binary proportion and 95% confidence interval for outcome measure ascertainment event rates.
Consent rate feasibility | 1 year
  Consent rate

OTHER OUTCOMES:
Leg and overall body strength at ICU awakening, ICU discharge, and hospital discharge | From study admission to approximately 5, 10, and 15 days, on average, respectively
  Manual muscle testing using the Medical Research Council (MRC) Scale. The patient exerts a force against the examiner's resistance. Each muscle is assessed on a 6-point MRC scale (0=no contraction; 5=contraction sustained against maximal resistance).
Quadriceps Leg Strength - hand held dynamometer at ICU awakening, ICU discharge, and hospital discharge | From study admission to approximately 5, 10, and 15 days, on average, respectively
  The patient exerts a force against a small strain gauge that fits in the examiner's hand. Force measured in Kg and in Newtons on a continuous scale.
Grip Strength - Hand grip dynamometer at ICU awakening, ICU discharge, and hospital discharge | From study admission to approximately 5, 10, and 15 days, on average, respectively
  Force measured in Kg. Force measured in Kg and in Newtons on a continuous scale.
Functional Status Scale for ICU at ICU awakening ICU, ICU discharge, and hospital discharge | From study admission to approximately 5, 10, and 15 days, on average, respectively
  The patient attempts 5 bed mobility/ transfer tasks: rolling, supine to sit, sitting at edge of be, transfer from sit to stand, ambulation. Each item assessed on a scale from 0 (unable to perform) to 7 (independent).
Katz Activities of Daily Living Scale at ICU awakening, ICU discharge, and hospital discharge | From study admission to approximately 5, 10, and 15 days, on average, respectively
  The patient's ability to complete 6 tasks: bathing, dressing, toileting, feeding, continence, and bed mobility. A rater assesses whether the patient is dependent or independent according to pre-specified criteria.
Physical Function Test for ICU at ICU awakening, ICU discharge, and hospital discharge | ICU awakening, ICU discharge, From study admission to approximately 5, 10, and 15 days, on average, respectively
  The patient completes 4 tasks: sit to stand, marching on the spot, repeated bilateral shoulder flexion, and muscle strength assessment (knee extension, shoulder flexion).
Patient-Specific Functional Scale at ICU awakening, ICU discharge, and hospital discharge | From study admission to approximately 5, 10, and 15 days, on average, respectively
  The patient rates their ability to complete a specific task on a scale from 0 (unable to perform activity) to 10 (able to perform activity at baseline level).

CONTACTS AND LOCATIONS:
Overall Officials: Michelle E Kho, PT, PhD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Intensive Care Unit, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Kho ME, Molloy AJ, McCaughan M, et al. TryCYCLE: Preliminary results of early in-bed cycling with mechanically ventilated patients. Crit Care Med 2014;43.
- [Derived] Kho ME, Molloy AJ, Clarke FJ, Ajami D, McCaughan M, Obrovac K, Murphy C, Camposilvan L, Herridge MS, Koo KK, Rudkowski J, Seely AJ, Zanni JM, Mourtzakis M, Piraino T, Cook DJ; Canadian Critical Care Trials Group. TryCYCLE: A Prospective Study of the Safety and Feasibility of Early In-Bed Cycling in Mechanically Ventilated Patients. PLoS One. 2016 Dec 28;11(12):e0167561. doi: 10.1371/journal.pone.0167561. eCollection 2016. PMID 28030555